CLINICAL TRIAL: NCT00903942
Title: A Modified Two Stage Phase II Study of Combination Abraxane and Radiation for Stage III Non-Small Cell Lung Cancer
Brief Title: Abraxane and RT for Non-Small Cell Lung Cancer (NSCLC)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: funding was withdrawn from Drug company
Sponsor: University of Rochester (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Yuhchyau Chen, MD, Ph.D, University of Rochester, Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RSRB00022397
Record Dates: First submitted 2009-05-15; First posted 2009-05-19 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Non-small Cell Lung Cancer, Stage III
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy; Taxes; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: radiation therapy — 1) PTV = CTV (GTV + 1.5-cm margins and the most adjacent nodal regions) + 0.5 cm margins to 5,040 cGy in 180 cGy daily fractions; and (2) Cone Down PTV = GTV +1.5 cm margins to 6,480 cGy.
Drug: Paclitaxel Protein-Bound, and CARBOPLATIN — Induction Chemotherapy Abraxane(260 mg/m2) / Carboplatin (AUC of 6) x one cycle Concurrent Chemotherapy(with radiation)--for first 3 pts--20 mg/m2 Abraxane, 3 times per week then for next group of 3 pts--30 mg/m2 Abraxane twice a week

SUMMARY:
For patients with stage III Lung Cancer, We propose one cycle chemotherapy using Abraxane and Carboplatin, followed by pulsed low-dose sensitizing Abraxane chemotherapy and daily Radiation. This will be followed by more hi-dose chemotherapy. We anticipate this regimen to target early distant microscopic spread by using one cycle of chemotherapy prior to radiation, and to achieve control of the disease in the lung by combining pulsed low-dose sensitizing Abraxane, with radiation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed NSCLC.
* Clinical or pathologic stage IIIA (T1-3N2M0, T3N1M0) and IIIB (Any T N3M0, T4 Any N M0) diseases according to the American Joint Committee of Cancer criteria.
* Patients with malignant pleural effusion will be excluded.
* The primary tumor must be radiographically measurable.
* Age > 18.
* Karnofsky performance status > 70 or Zubrod PS 0 or 1.
* FEV1 sufficient for patients to tolerate radiation therapy, which is at the discretion of the radiation oncologist, usually > 800 ml, but may be higher or lower depending on the volume of radiotherapy portal, which is a variable of the tumor extent.
* WBC > 3000; platelet count > 100,000; absolute neutrophil counts > 1,500; HGB > 9.0 g/dl, serum creatinine < 1.5 mg/dl or creatinine clearance > 60 ml/min. Laboratory values must be obtained < 4 weeks prior to registration.
* Patients with equivocal enlargement of adrenal gland(s) on CT scan, or a few equivocal regional or distant lesions on any imaging studies need further imaging study (PET, bone scan, or others) or biopsy to rule out distant metastasis.
* Patients must have adequate liver functions: AST and ALT < 2.5 x upper limit of normal, alkaline phosphatase < 2.5 x upper limit of normal, unless bone metastasis is present in the absence of liver metastasis. Bilirubin <1.5 mg/dL.
* Pre-existing neuropathy must not be worse than grade I.
* A signed informed consent.
* Normal organ function including EKG findings deemed acceptable for chemotherapy by the medical oncologist.

Exclusion Criteria:

* Patients with distant metastasis (stage IV disease).
* Patients without measurable disease.
* Patients with medical contraindication to chemotherapy or radiotherapy.
* Patients with myocardial infarction within the preceding 6 months or symptomatic heart disease, including angina, congestive heart failure, uncontrolled arrhythmia.
* Patients with bilirubin elevated above institutional upper limit of normal (ULN) must be excluded.
* Women who are pregnant or breastfeeding are not eligible.
* Other serious illnesses or medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-03; Primary Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
To assess feasibility of one cycle induction chemotherapy of Abraxane plus Carboplatin followed by low-dose sensitizing Abraxane and radiation followed by consolidation Abraxane and carboplatin for stage III NSCLC. | 4 years

SECONDARY OUTCOMES:
To estimate the local tumor response rate | 4 years
To estimate 2-year in-field tumor control. | 6 year
To estimate 2-year disease free survival (DFS). | 6 years
To estimate 2-year overall survival (OS). | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Yuhchyau Chen, MD,PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Medical Center, Rochester, New York, United States